CLINICAL TRIAL: NCT03489239
Title: Long-term Study to Observe Safety and Efficacy of TAF in Patients With Chronic Hepatitis B
Brief Title: Entecavir to TAF Switch
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11729
Record Dates: First submitted 2018-03-14; First posted 2018-04-05 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): SingleArm: TAF 25 mg
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — subjects switching from Entecavir to single arm TAF 25mg
  Other Names: TAF

SUMMARY:
A research study to observe the safety, efficacy and tolerability of switching from Entecavir (ETV) to Tenofovir Alafenamide TAF in patients with chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

* Subjects, adult male and female ≥18 years of age with chronic hepatitis B with or without compensated cirrhosis
* Maintained on Entecavir for a minimum of 48 weeks
* Viral suppression (HBV DNA <20 IU/mL) for a minimum of 12 weeks prior to entry are eligible for this study.
* Estimated creatinine clearance ≥ 50 ml/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the baseline evaluation.

Exclusion Criteria:

* Subjects with known poor or non-compliance
* Subjects with co-infection with HCV or HIV subjects with decompensated cirrhosis and HCC will be excluded to participate in the study.
* Pregnant women and those who wish to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-16 (Estimated)

PRIMARY OUTCOMES:
Results of viral Hepatitis B DNA to be <20 IU/mL | 48 weeks
  The proportion of subjects with plasma HBV DNA levels below 20 IU/mL at week 48.

SECONDARY OUTCOMES:
Complete viral suppression at study completion | 96 Weeks
  The proportion of subjects with complete viral suppression, i.e., plasma HBV DNA level below 20 IU/mL at Week 96.
Positive eGFR changes at study completion compared to Baseline visit | 96 weeks
  Change in eGFR from baseline to Week 96
Improved Bone Mass Density at study completion | 96 weeks
  % change from baseline in BMD at the hip and lumbar spine at Week 96.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States